CLINICAL TRIAL: NCT02138188
Title: Psychological Aspects and Continuous Subcutaneous Insulin Infusion in Type 1 Diabetic Adults.
Brief Title: Psychological Aspects and Insulin Pump Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Maddalena Trombetta, MD, PhD, Universita di Verona
Other Study IDs: ISP-DT1-ITA13 (CE-2393)
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- T1D patients on CSII: Patients affected by Type 1 Diabetes on insulin pump therapy

SUMMARY:
The Continuous Subcutaneous Insulin Infusion (CSII) might have an impact on psychological distress and some psychological factors might be predictors of metabolic control; however, very few studies conducted so far were specifically focused on the psychological aspects of CSII therapy in adults affected by T1DM.

DETAILED DESCRIPTION:
The aim of this project is to study the psychological effect of Continuous Subcutaneous Insulin Infusion (CSII) in a cohort of type 1 diabetic patients and to explore the influence of psychological factors (coping style, locus of control, self-efficacy) on glycaemic control. A sample of 36 type 1 diabetic patients will be recruited at Endocrinology, Diabetes and Metabolism Division of Verona City Hospital.

Among T1DM patients routinely followed by our Institution the study will be proposed to those starting the CSII therapy based on the inclusion and exclusion criteria.

Each study participants will provide a written informed consent and will undergo a set of 4 psychological evaluation assessing depression, anxiety, self-efficacy, perceived interference caused by diabetes, family support, locus of control and coping strategies on top of routine medical examination and laboratory testing for outcome measures at baseline and after 6, 12 and 24 months after study entry.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes
* Transition to CSII
* Age >18 years

Exclusion Criteria:

* Current schizophrenia/ psychotic disorders, bipolar disorders, addictive disorders, personality disorders
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient setting
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline glycosylated haemoglobin (HbA1c) at 6th, 12th and 24th months after transition to CSII. | Baseline, 6, 12 and 24 months
  Glycosylated haemoglobin (HbA1c) is a lab test that shows the average level of blood glucose over the previous 3 months. HbA1c is used in the present study as measure of the glycaemic control: it will be assessed at baseline, after 6, 12 and 24 months.

SECONDARY OUTCOMES:
Change from baseline glucose variability as measured by standard deviation (SD) and coefficient of variation (CV) of capillary blood glucose test [mg/dL] at 6th, 12th and 24th months after transition to CSII. | Baseline, 6, 12, 24 months
  SD and CV will be calculated from daily measurements of at least 3 capillary blood glucose measurements representative of pre- and post-meal glucose excursion over the entire day.
Change from baseline glucose variability as measured by the Low Blood Glucose Index (%LBGI) at 6th, 12th and 24th months after transition to CSII. | Baseline, 6, 12, 24 months
  The LBGI is a validated percentage index of frequency and amplitude of glucose excursions below a conventional glucose threshold set at 6.25 mmol/L and allows the normalization of non-Gaussian distributions of both capillary and interstitial blood glucose measurements collected over a pre-determined time frame.
Change from baseline glucose variability as measured by High Blood Glucose Index (%HBGI) at 6th, 12th and 24th months after transition to CSII. | Baseline, 6, 12, 24 months
  The HBGI is a validated percentage index of frequency and amplitude of glucose excursions over a conventional glucose threshold set at 6.25 mmol/L, as previously described.
Change from baseline depressive symptoms at 6th,12th and 24th months (BDI-II score) | Baseline, 6, 12, 24 months
  The Beck Depression Inventory II is a 21-item questionnaire developed to assess the intensity of depression as defined by the Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition (DSM-IV). The BDI-II items include cognitive symptoms such as sadness and pessimism, affective symptoms such as loss of pleasure and loss of interest, somatic symptoms such as loss of energy, appetite changes and changes in sleep pattern. The BDI-II is calculated by summing the ratings for the 21 items. The 4-point scale ranges from 0 to 3 for each item. The maximum total score is 63. The measurement of outcome variables will be conducted 6, 12 and 24 months after transition to CSII.
  The difference of the BDI-II scores among baseline, at 6,12 and 24 months will be also calculated.
Change from baseline anxiety symptoms at 6th,12th and 24th months (BAI score) | Baseline, 6, 12, 24 months
  The Beck Anxiety Inventory is a 21- item questionnaire developed to assess the severity of anxiety by describing its emotional, physiological and cognitive symptoms. The 4-point scale of BAI score ranges from 0 to 3 for each item, with a maximum total score of 63. Outcome variables will be evaluated at 6, 12 and 24 months after transition to CSII. The difference of the BAI scores among baseline, 6, 12 and 24 months will be also calculated.
Change from baseline general perceptions of diabetes at 6th, 12th and 24th months (MDQ Section 1 score) | Baseline, 6, 12, 24 months
  The Multidimensional Diabetes Questionnaire (MDQ) was designed to provide a comprehensive assessment of diabetes-related cognitive and social factors. It includes 41 items subcategorized in three sections. The first section assesses the general perceptions of diabetes and related social support. It is comprised of three scales. These scales targets:
  perceived interference caused by diabetes to daily activities, work and social activities (9 items); perceived severity of diabetes (3 items); perceived diabetes-related social support from a significant other such as family, friends and health professionals (4 items).
  Responses were rated on 7-point rating scales (from 0 to 6), with higher scores indicating higher levels of perceived interference, social support and severity.
Change from baseline family support at 6th, 12th and 24th months (MDQ section II score) | Baseline, 6, 12 and 24 months
  This section of the MDQ measures social incentives in relation to self-care activities. The scales included in this section were designed to measure the frequency of positive reinforcing behaviour (8 items) and the frequency of non supportive behaviours (4 items). Subjects recorded their responses on 7-point Likert scales (from 0 to 6) with higher scores indicating higher levels of positive and negative reinforcement behaviours.
Change from baseline Diabetes Self-Efficacy at 6th, 12th and 24th months (MDQ section III score) | Baseline, 6, 12, 24 months
  This section of the MDQ is used to assess self-efficacy expectancies (7 items) and outcome expectancies (6 items). The self-efficacy scale measured patients' confidence in their ability to perform behaviors specific to the diabetes self-care activities. Responses were rated on a 0 to 100 rating scale. The outcome expectancies scale assessed patients' perceptions of the effect of diabetes self-care behaviors on metabolic control. Responses were rated on a 0 to 100 rating scale.
Determination of Health Locus of Control (MHLC) at Baseline | Baseline
  The multidimensional Health Locus of Control Scale consists of three subscale with six items each. The three subscales are: Internal Health Locus of Control (IHLC), Powerful Others Externality (PHLC), Chance Health Locus of Control (CHLC).
Measures of Coping Strategies at Baseline | Baseline
  Coping strategies will be measured with the Coping Orientation to Problems Experienced-New Italian Version (COPE-NVI). The instrument is a multidimensional 60-items coping inventory to assess the different ways in which people respond to stress and it was developed to assess a broad range of coping responses.

CONTACTS AND LOCATIONS:
Overall Officials: Maddalena Trombetta, MD Phd, Principal Investigator — AOUI Verona
Locations (1):
- Division of Endocrinology, Diabetes and Metabolism-Department of Medicine-AOUI Verona, Verona, Italy